CLINICAL TRIAL: NCT01282541
Title: Determination of the Optimum Delivery Route for the Intraglandular Administration of Botulinum Toxin A in Patients With Refractory Epiphora
Brief Title: Determination of the Optimum Delivery Route for Botulinum Toxin A in Patients With Epiphora
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merbs, Shannath, M.D., Ph.D. (Individual)
Responsible Party: Principal Investigator, Shannath Merbs, M.D., Ph.D., Associate Professor of Ophthalmology and Oncology, Merbs, Shannath, M.D., Ph.D.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00025405
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Epiphora
Keywords: Tearing, Epiphora, Botulinum Toxin A
MeSH Terms: conditions — Lacrimal Apparatus Diseases; Lacerations | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transconjunctival (Active Comparator)
  Interventions: Drug: Botulinum Toxin Type A
- Transcutaneous (Active Comparator)
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A — 100 units/2ml 0.9% sodium chloride, 5 units delivered transconjunctivally into the palpebral lobe of the lacrimal gland once
  Other Names: Botox
  Arms: Transconjunctival
Drug: Botulinum Toxin Type A — 100 units/2ml 0.9% sodium chloride, 5 units delivered transcutaneously into the orbital lobe of the lacrimal gland once
  Other Names: Botox
  Arms: Transcutaneous

SUMMARY:
Epiphora or excessive tearing is a significant disability for many affected patients diminishing their quality of life. There is a growing consensus that injection of Botulinum Toxin A (BTX-A) into the lacrimal gland provides relief in patients with hyperlacrimation secondary to aberrant regeneration of the 7th nerve, and limited evidence that it might help to reduce normal tear production in patients with epiphora from anatomic or functional outflow obstructions. BTX-A has been injected both transconjunctivally into the palpebral lobe of the lacrimal gland and transcutaneously into the orbital lobe. Both delivery routes have been successful in symptom relief with minimal complications. However, the effectiveness of transconjunctival versus transcutaneous injections has not been systematically compared. Also, whether the incidence of side effects is related to the dosage, concentration, or location of injection is unknown and has also not been systematically studied. The investigators plan to conduct a randomized clinical trial in patients with functional tearing comparing the transcutaneous delivery route of BTX-A to the transconjunctival delivery route (the most common route described in the literature). The investigators will also compare the side effect profile of each delivery route.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* ability to give informed consent
* symptoms of epiphora in the setting of either a patent lacrimal outflow system or an obstructed outflow system for which the patient does not desire surgical therapy or is a poor surgical candidate

Exclusion Criteria:

* pregnancy
* ocular motility abnormalities
* prior ptosis, and/or strabismus surgery
* more than 2 mm of pre-existing ptosis
* inability to give informed consent
* history of a bleeding disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Comparison of 1-minute Schirmer's test with and without anesthesia between treatment groups at baseline and follow up | 24 weeks

SECONDARY OUTCOMES:
Comparison of side effect between each treatment group | 24 weeks
Comparison of average score on epiphora severity scale between groups of interest at baseline and follow-up | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shannath Merbs, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States